CLINICAL TRIAL: NCT05574621
Title: Comparison of Inflammatory Markers, Oxidative Stress, Platelet Activation and Autophagy Between Internal Thoracic Artery and Left Anterior Descending Artery in Patients Subjected to Off-pump Surgical Myocardial Revascularization
Brief Title: ITA Vs LAD; Evaluation of Inflammatory Burden in OP-CABG Patients
Status: Completed | Type: Observational
Sponsor: Cardiochirurgia E.H. (Other)
Collaborators: University of Roma La Sapienza (Other); Andrea Salica (Unknown); Francesco Giosuè Irace (Unknown)
Responsible Party: Sponsor
Other Study IDs: EH2021-01
Record Dates: First submitted 2022-10-01; First posted 2022-10-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease; Atherosclerosis; Inflammation
Keywords: coronary artery bypass graft; coronary revascularization
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Atherosclerosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collected for internal thoracic artery and left descending artery
Oversight: Data Monitoring Committee: No

SUMMARY:
Introduction. Ischemic cardiomyopathy is one of the death leading causes in industrialized countries. Up-to-date ESC guidelines recommend a surgical approach (coronary by pass graft) in patients with multivessel coronaropathy, with involvement of left main (LM) or proximal left anterior descending (LAD) artery. In any case, is recommended the use of the internal thoracic artery (ITA) as conduct of choice.

In consideration of the very strong evidence supporting the use of ITA, the study objective is to analyze and compare some blood markers collected from ITA blood vs. LAD blood, with the purpose of better understanding the technique benefits from a biological point of view, being the hemodynamic one already evident.

Methods. Forty patients scheduled for coronary bypass graft (CABG) surgery at the Cardiac Surgery Unit of European Hospital of Rome will be enrolled. Patients which intervention includes off-pump ITA-LAD anastomosis will be included. For each patient blood sample from ITA and LAD will be collected. On those samples, polymorphonuclear leukocytes and platelets activity, endothelial dysfunction, oxidative stress and inflammatory burden will be analysed. In patients in which a pre-operative coronary CT scan is available, findings will be correlated with atherosclerotic plaque morphology.

Expected results. Diseased LAD's blood will have a deranged markers profile compared with ITA's, with augmented inflammatory burden, reduce NO availability and increased platelet activation. In the patients subgroup with available coronary CT scan will be possible to esteem the effective blood mixing and speculate on a possible pharmacological effect of CABG, in terms of dilution of inflammatory burden in the target vessel.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled coronary bypass surgery
* Off-pump procedure
* ITA-LAD anastomosis

Exclusion Criteria:

* STEMI in the last month
* LVEF > 30%
* LAD chronic occlusion
* Acute or chronic inflammatory diseases
* Immunologic or rheumatic diseases
* Oncologic condition (present or in the last 3 years)
* Active infections

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited among the all-comers surgical candidates at European Hospital of Rome, which includes out patient clinic, internal transfers from cardiology unit, urgent transfers from other regional hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory burden | through study completion, an average of 6 months
  Serum inflammatory cytokines, evaluated through enzyme-linked immunosorbent assays (ELISA)

SECONDARY OUTCOMES:
Oxidative stress | through study completion, an average of 6 months
  soluble NOX-derived peptide evaluated through ELISA; H2O2 evaluated with colorimetric test

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy